CLINICAL TRIAL: NCT01489423
Title: Correlative Analyses of Specimens From Eastern Cooperative Group Study E1608
Brief Title: Tissue and Blood Biomarkers From Patients With Stage III or Stage IV Melanoma Treated With Ipilimumab With or Without Sargramostim
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000718014; ECOG-E1608T1
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IIIC melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — In Situ Hybridization; Polymerase Chain Reaction; Enzyme-Linked Immunosorbent Assay; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: RNA analysis
Genetic: in situ hybridization
Genetic: polymerase chain reaction
Other: enzyme-linked immunosorbent assay
Other: flow cytometry
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue and blood in the laboratory from patients treated with ipilimumab with or without sargramostim may help doctors learn more about the effects of ipilimumab and sargramostim on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research trial studies tissue and blood biomarkers in patients with stage III melanoma or stage IV melanoma treated with ipilimumab with or without sargramostim.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the pathology of primary melanomas, melanoma metastases, and post-treatment melanoma metastases in relation to clinical outcomes for patients receiving ipilimumab plus sargramostim (GM-CSF) and patients receiving ipilimumab alone.
* To determine the effects of the addition of systemic GM-CSF to ipilimumab on effector immune function in patients with metastatic melanoma.
* To determine the effects of the addition of systemic GM-CSF to ipilimumab on regulatory immune function in patients with metastatic melanoma.
* To determine the effects of the addition of systemic GM-CSF to ipilimumab on anti-tumor humoral immunity in patients with metastatic melanoma.

OUTLINE: Serum, peripheral blood mononuclear cells, and tumor tissue (from primary tumor and post-treatment biopsies) samples are analyzed for biomarkers predictive of clinical outcomes, immune function, and anti-tumor humoral immunity by IHC, RT-PCR, flow cytometry, ELISPOT assays, and ELISA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of measurable unresectable stage III or stage IV melanoma
* Treated with ipilimumab with or without sargramostim on clinical trial ECOG-E1608
* Primary tumor tissue and optional post-treatment biopsies of tumors from easily accessible tissues

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients who participated in E1608 and provided samples for research.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2013-04-26 (Actual); Primary Completion 2013-05-26 (Actual); Study Completion 2013-05-26 (Actual)

PRIMARY OUTCOMES:
Primary brisk lymphocytic infiltrates associated with better outcomes (overall survival, progression-free survival, and clinical response) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute